CLINICAL TRIAL: NCT06355128
Title: A Cross-sectional Study of Ocular Manifestations During the Covid-19 Pandemic in Hubei Province
Status: Active, not recruiting | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Collaborators: Qichun People's Hospital (Unknown)
Responsible Party: Principal Investigator, Min Ke, Director of Ophthalmology, Zhongnan Hospital
Other Study IDs: 20240307
Record Dates: First submitted 2024-03-21; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: COVID-19; Ocular Surface Disease
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- the pandemic period (Phase A): the pandemic period (Phase A)
  Interventions: Other: NOT
- the prevention and control periods (Phase B: November 7, 2022 to December 6, 2022 ).: the prevention and control periods (Phase B: November 7, 2022 to December 6, 2022 and Phase C: December 7, 2021 to January 6, 2022).
  Interventions: Other: NOT
- the prevention and control periods (Phase C: December 7, 2021 to January 6, 2022).: the prevention and control periods (Phase B: November 7, 2022 to December 6, 2022 and Phase C: December 7, 2021 to January 6, 2022).
  Interventions: Other: NOT

INTERVENTIONS:
Other: NOT — NOT

SUMMARY:
To investigate the clinical features of ocular manifestations during the novel coronavirus pneumonia pandemic in Hubei at the end of 2022

DETAILED DESCRIPTION:
During late 2022 COVID-19 pandemic ocular discomforts were common in people with mild systemic symptoms, but most resolve on their own without any treatment. The disease spectrum of ophthalmology outpatient clinics is affected by the COVID-19 pandemic. In our study, we observed that the incidence of keratitis and acute angle-closure glaucoma in Phase A was significantly higher than that in Phase B and C.

ELIGIBILITY:
Inclusion Criteria:

* 1. 2022.12.7 to 2023.2.6 People surveyed by wechat Questionnaire Star 2. 2021.12.7 to 2022.1.6 and 2022.11.7 to 2023.1.6 Patients who received ophthalmology treatment in Zhongnan Hospital of Wuhan University and Qichun People's Hospital

Exclusion Criteria:

* 1. currently hospitalized patients. 2. severe patients. 3. Incomplete information. 4. cannot be contacted by telephone. 5. Refuse questionnaire survey. 6.The electronic medical record information is incomplete. 7. Those who do not go to the ophthalmic clinic after registration. 8.severe patients. 9. Cannot be contacted by phone.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: People from Hubei Province, China
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-18 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Questionnaire data were collected and statistically analyzed. | 1/4/2024-30/4/2024
  Information on demographic characteristics, COVID-19 pathogen test results, Covid-19 related systemic symptoms, ocular symptoms and eye discomfort medication was collected from questionnaires during the pandemic period (Phase A: December 7, 2022 to January 6, 2023, 1968 patients). Electronic medical records in the ophthalmic outpatient department of Zhongnan Hospital of Wuhan University and its medical union hospital- Qichun County People's Hospital were extracted during the pandemic period (Phase A) and the prevention and control periods (Phase B: November 7, 2022 to December 6, 2022 and Phase C: December 7, 2021 to January 6, 2022). The demographic, epidemiological, and clinical information of patients were compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China